CLINICAL TRIAL: NCT06393218
Title: The Impact of Diaphragm Training on Dysphagia in Bulbar Palsy After Ischemic Stroke: A Randomized Controlled Study
Brief Title: The Impact of Diaphragm Training on Dysphagia in Bulbar Palsy After Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEJI-Zhenqiu
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Bulbar Palsy
MeSH Terms: conditions — Bulbar Palsy, Progressive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine rehabilitation+Diaphragm Training (Experimental): Study lasts 15 days for each patient. The patients were given comprehensive rehabilitation therapy. The observation group was provided the support of enteral nutrition by Intermittent Oro-esophageal Tube Feeding. Diaphragm Training will be given twice a day and 30min per time.
  Interventions: Device: Intermittent Oro-esophageal Tube Feeding; Behavioral: Diaphragm Training; Behavioral: Routine rehabilitation
- Routine rehabilitation (Active Comparator): Study lasts 15 days for each patient. The patients were given comprehensive rehabilitation therapy. The observation group was provided the support of enteral nutrition by Intermittent Oro-esophageal Tube Feeding.
  Interventions: Device: Intermittent Oro-esophageal Tube Feeding; Behavioral: Routine rehabilitation

INTERVENTIONS:
Device: Intermittent Oro-esophageal Tube Feeding — Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
Behavioral: Diaphragm Training — Diaphragm training includes both active and passive methods. Passive training involves placing weights on the participant's abdomen to provide resistance during breathing. Active training involves instructing participants to practice diaphragmatic breathing techniques.
  Arms: Routine rehabilitation+Diaphragm Training
Behavioral: Routine rehabilitation — Including： Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.

SUMMARY:
This was a prospective multicenter study. the patients after stroke with were randomly divided into the observation group and the control group. All patients were given comprehensive rehabilitation therapy. During the treatment, enteral nutrition support was provided for the two groups by Intermittent Oro-esophageal tube feeding. The observation group will be given Diaphragm Training Nutritional status, dysphagia, quality of life and depression before and after treatment were compared.

DETAILED DESCRIPTION:
Dysphagia in patients after stroke continues to be a challenge. This was a prospective multicenter study. the patients after stroke with were randomly divided into the observation group and the control group. All patients were given comprehensive rehabilitation therapy. During the treatment, enteral nutrition support was provided for the two groups by Intermittent Oro-esophageal tube feeding. The observation group will be given Diaphragm Training Nutritional status, dysphagia, quality of life and depression before and after treatment were compared.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* meeting the diagnostic criteria of Bulbar Palsy After Ischemic Stroke;
* any degree of dysphagia at admission;
* steady vital signs, without severe cognitive impairment or sensory aphasia, able to cooperate with the assessment.
* clear mind.

Exclusion Criteria:

* complicated with other neurological diseases;
* damaged mucosa or incomplete structure in nasopharynx;
* tracheostomy tube plugged;
* unfeasible to the support of parenteral nutrition;
* simultaneously suffering from liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | Day 1 and day 15
  The Penetration-Aspiration Scale was conducted under video fluoroscopic swallowing study. The scale is a standardized tool used to assess the safety of swallowing. The scale was developed to evaluate the entry of material into the airway (penetration) and the subsequent passage of material below the vocal folds (aspiration) during swallowing. The scale ranges from 1 to 8, with each level representing different degrees of penetration or aspiration.

SECONDARY OUTCOMES:
Functional Oral Intake Scale | Day 1 and day 15
  The scale reflects the patient's oral intake. Studies have shown that this scale can also serve as an independent measure of intake for post-stroke dysphagia patients. The scale is divided into 7 levels, with the level positively correlated with swallowing function. Level 7 indicates normal swallowing function.
Dysphagia Handicap Index | Day 1 and day 15
  Dysphagia Handicap Index is a self-reported questionnaire used to assess the impact of dysphagia on an individual's quality of life. It typically consists of multiple questions related to the physical, functional, and emotional aspects of swallowing difficulties. The total score range varies between 0 and 100. A higher score indicates a greater perceived impact of dysphagia on the individual's quality of life.